CLINICAL TRIAL: NCT07097506
Title: Effect of Ketone Esters on Liver Fat and Metabolic Function in Adolescents With Obesity and MASLD
Brief Title: Effect of Ketone Esters on Liver Fat Content and Metabolic Function
Acronym: JV
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Children's Discovery Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202503064
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: MASLD - Metabolic Dysfunction-Associated Steatotic Liver Disease; Obesity; Overweight (BMI > 25)
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, placebo controlled study design
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): 25 g Placebo per day for approximately 6-weeks
  Interventions: Other: Placebo
- C8 ketone di-ester (Experimental): 25 g C8 ketone di-ester per day for approximately 6-weeks
  Interventions: Drug: bis-octanoyl (R)-1,3-butanediol (C8 ketone di-ester)

INTERVENTIONS:
Drug: bis-octanoyl (R)-1,3-butanediol (C8 ketone di-ester) — 25 g C8 ketone di-ester taken daily for approximately 6-weeks
  Other Names: Qitone
  Arms: C8 ketone di-ester
Other: Placebo — 25 g Placebo taken daily for approximately 6-weeks
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to determine whether ingestion of a ketone ester drink helps improve liver health and blood glucose control. Ketones are a type of energy source made by the body during times of weight loss, low carbohydrate intake and starvation.

People enrolled in this study will be randomly assigned (by chance, like the flip of a coin) to one of two groups:

Group 1: Ketone ester drink consumed daily for 6 weeks. Group 2: Placebo drink consumed daily for 6 weeks.

DETAILED DESCRIPTION:
Metabolic dysfunction-associated steatotic liver disease (MASLD) is a common complication of obesity and is associated with multiorgan insulin resistance, dyslipidemia (high plasma triglyceride and low HDL cholesterol concentrations), and an increased risk of diabetes and coronary heart disease. The prevalence of MASLD continues to rise dramatically in children and adolescents, with approximately 13 to 19% of adolescents and young adults in the United States estimated to have hepatic steatosis (elevated amount of fat in the liver), the hallmark feature of MASLD. Evidence is emerging that increasing blood ketone concentrations can markedly improve hepatic steatosis, insulin sensitivity, and blood glucose in rodent models of obesity.

Ketones are produced by the liver from fatty acid metabolism; increased ketone production is observed during fasting or very-low carbohydrate (ketogenic) diet consumption when plasma nonesterified fatty acid concentrations are high and glucose concentrations are low. Circulating ketone concentrations can also be increased by exogenous ketone administration. Ketogenic diets ameliorate hepatic steatosis in adults with MASLD. Whether exogenous ketone administration affects hepatic steatosis in adolescents with MASLD is not known. However, several studies have found exogenous ketone administration improves blood glucose control in people, suggesting that exogenous ketones could also reduce intrahepatic triglyceride (IHTG) content.

The therapeutic use of ketone drinks has been limited by poor palatability and the high sodium content of ketone salts. To overcome these limitations, ketone esters have recently been developed, including bis-octanoyl (R)-1,3-butanediol (C8 ketone di-ester), which is hydrolyzed in the intestine to generate the ketone precursors octanoic acid and (R)-1,3-butanediol, which are then converted to beta-hydroxybutyrate by the liver. These ketone precursors are palatable, do not contain sodium, and have been shown to increase plasma ketone concentrations. The purpose of the present study is to conduct a randomized double blind, placebo-controlled 6-week trial to assess the effect of C8 ketone di-ester supplementation (25 g/day) on IHTG content and blood glucose control (insulin sensitivity, beta-cell function, glucose tolerance) in 40 adolescents with obesity and MASLD.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥18 and ≤25 years;
* BMI 25.0 - 44.9 kg/m2;
* Intrahepatic triglyceride content >5% assessed by using magnetic resonance imaging-proton density fat fraction (MRI-PDFF).

Exclusion Criteria:

* HbA1C ≥6.5%;
* taking dietary supplements or medications known to affect our study outcomes including corticosteroids and other drugs associated with steatosis (metformin use will be allowable if participants have taken a stable dose for at least 3 months without any gastrointestinal-related symptoms);
* active eating disorder, any anaphylactic food allergy and/or consuming a very-low-carbohydrate (<50 g/day) diet;
* Fibroscan controlled attenuation parameter (CAP) score <240 dB/m assessed within last 2 months before entering the study;
* recent (<2 months) history of moderate-severe nausea, vomiting, diarrhea, or other significant gastrointestinal symptoms;
* consume tobacco products, excessive alcohol (females: >14 drinks/week; males: >21 drinks/week), or illegal drugs determined by medical history;
* evidence of significant active organ system dysfunction, liver disease other than MASLD (e.g., Wilson disease, viral hepatitis, inborn errors of metabolism, or alpha-1 antitrypsin deficiency) or cirrhosis as a results of any condition or disease;
* have had bariatric surgery or plan to have endoscopic or bariatric surgery therapy for obesity;
* have undergone organ transplantation;
* have HIV and any other type of congenital or acquired lipodystrophy;
* unwilling or unable to provide informed consent;
* major psychiatric illness;
* metal implants that are not MRI-compatible;
* pregnancy, as determined by a urine HCG screening test assessed performed at all screening, baseline testing, and follow-up visits. In addition, male and female participants of reproductive and childbearing age who wish to enroll will be required to agree to use contraception throughout the study period, and for 30 days after the last dose of C8 ketone di-ester;
* female participants who are currently lactating;
* Structured exercise: ≥75 min/wk of vigorous exercise (e.g., jogging, activity that causes heavy breathing and sweating) or ≥200 min/wk of low intensity physical activity (e.g., brisk walking);
* Unstable weight (>3% change during the last 2 months before entering the study);
* Anemia (hemoglobin <10.5 g/dL in females and <11.0 g/dL in males);
* Unable or unwilling to follow the study protocol or who, for any reason, is considered an inappropriate candidate for the study by the research team.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-26 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Intrahepatic triglyceride content | Before and at the end of treatment at 6-weeks
  Intrahepatic triglyceride content will be assessed by magnetic resonance imagining (MRI)
Change in insulin sensitivity | Before and at the end of treatment at 6-weeks
  Whole-body insulin sensitivity will be assessed by using the hyperinsulinemic-euglycemic clamp procedure

SECONDARY OUTCOMES:
Change in β-cell function | Before and at the end of treatment at 6-weeks
  β-cell function will be assessed from a modified oral glucose tolerance test
Change in glycemic control | Before and at the end of treatment at 6-weeks
  Glycemic control will be assessed by using an oral glucose tolerance test

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Klein, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States